CLINICAL TRIAL: NCT06889883
Title: Development and Validation of a Blood Test for Early Diagnosis of Colorectal Cancer Based on Molecular Markers and Risk Factors Identified With Artificial Intelligence Tools
Brief Title: Development and Validation of a Blood Test for Early Diagnosis of Colorectal Cancer
Acronym: ColoDix
Status: Recruiting | Type: Observational
Sponsor: ADVANCED MARKER DISCOVERY S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMD-CCR-2022-02
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Carcinoma; Advanced Adenomas (AA)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy: Individual with no findings or findings not related to neoplasia on colonoscopy
- Advanced Adenoma: Patient diagnosed with advanced adenoma by colonoscopy and confirmed by histology result
- Colorectal Cancer: Patient diagnosed with colorectal cancer by colonoscopy and confirmed by histology result

SUMMARY:
This is a prospective, multicenter, case-control study. The aim is to develop an optimized algorithm by combining the levels of molecular markers in plasma together with risk factors for developing colorectal cancer and clinical data of patients diagnosed with CRC or AA and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who are able to understand the participant information and sign the informed consent.
* Patients who are going to undergo colonoscopy or surgical resection for tumor (CRC).

Exclusion Criteria:

* Patients who had developed any type of cancer in the 5 years prior to their participation in this study.
* Patients who have received previous chemotherapy or radiotherapy.
* Patients diagnosed with non-advanced adenomas, serrated polyps, Familial Adenomatous Polyposis or Lynch Syndrome.
* Patients with inadequate bowel preparation for colonoscopy.
* Patients who have undergone colonoscopy/polipectomy in the previous 5 years.
* Patients with hemolyzed plasma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study involves the recruitment of 510 patients as part of a case-control study. Patients who are going to undergo colonoscopy or who are going to undergo surgery for resection of a CRC already diagnosed will be included. They can be symptomatic or asymptomatic, ambulatory, hospitalized or consecutive patients in the Endoscopy Unit.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Validation | 36 months
  To clinically validate the diagnostic capability of the algorithm for early detection of CRC and AA that combines molecular markers and risk factors

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario de Cruces, Bilbao, Basque Country
  - Policlinica Gipuzkoa Hospital, Donostia / San Sebastian, Basque Country
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Sant Rafael, Barcelona, Catalonia
  - Hospital Universitario Vall d' Hebron, Barcelona, Catalonia
  - MD Anderson Cancer Centre, Madrid, Madrid
  - Hospital Centro Médico de Asturias, Oviedo, Principality of Asturias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herreros-Villanueva M, Duran-Sanchon S, Martin AC, Perez-Palacios R, Vila-Navarro E, Marcuello M, Diaz-Centeno M, Cubiella J, Diez MS, Bujanda L, Lanas A, Jover R, Hernandez V, Quintero E, Jose Lozano J, Garcia-Cougil M, Martinez-Arranz I, Castells A, Gironella M, Arroyo R. Plasma MicroRNA Signature Validation for Early Detection of Colorectal Cancer. Clin Transl Gastroenterol. 2019 Jan;10(1):e00003. doi: 10.14309/ctg.0000000000000003. PMID 30702491
- [Background] Giraldez MD, Lozano JJ, Ramirez G, Hijona E, Bujanda L, Castells A, Gironella M. Circulating microRNAs as biomarkers of colorectal cancer: results from a genome-wide profiling and validation study. Clin Gastroenterol Hepatol. 2013 Jun;11(6):681-8.e3. doi: 10.1016/j.cgh.2012.12.009. Epub 2012 Dec 23. PMID 23267864
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338